CLINICAL TRIAL: NCT01789645
Title: Efficacy of Conservative Versus Surgical Therapy for Carpal Tunnel Syndrome: a Randomised Clinical Trial
Brief Title: Physical Therapy in Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Collaborators: Hospital Universitario Fundación Alcorcón (Other)
Responsible Party: Principal Investigator, César Fernández-de-las-Peñas, Professor, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI01223
Record Dates: First submitted 2013-02-06; First posted 2013-02-12 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal tunnel; Physical therapy; Surgery; Efficacy
MeSH Terms: conditions — Carpal Tunnel Syndrome; Median Neuropathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conservative group (Experimental): The conservative group will received 3 treatment sessions of physical therapy based on neuromodulation of nociceptive processing of 30 minutes of duration, once per week.
  Interventions: Other: Conservative group
- Surgical group (Active Comparator): The surgical group will receive the surgical procedure consisting of the decompression and release of the median nerve at the carpal tunnel performed by an experienced surgeon according to standardized protocols.
  Interventions: Procedure: Surgical group

INTERVENTIONS:
Other: Conservative group — The conservative group will received 3 treatment sessions of physical therapy based on neuromodulation of nociceptive processing of 30 minutes of duration, once per week.
  Arms: Conservative group
Procedure: Surgical group — The surgical group will receive the surgical procedure consisting of the decompression and release of the median nerve at the carpal tunnel performed by an experienced surgeon according to standardized protocols.
  Arms: Surgical group

SUMMARY:
It is a randomized clinical trial comparing surgical and conservative (physical therapy) treatments for women with carpal tunnel syndrome (CTS). The purpose of the study is to determine the efficacy of physical therapy versus endoscopic surgery in pain and disability in women with carpal tunnel syndrome at medium and long-term follow-up periods. We hypothesized that proper physical therapy approach can be equally effective than surgical intervention for improving pain and function in patients with carpal tunnel syndrome.

DETAILED DESCRIPTION:
Scientific evidence for the management of CTS has exhibited conflicting results. The Cochrane review concluded that surgical treatment relieves symptoms significantly better than splinting but further research is needed. A systematic review focused on physical therapy for the management of CTS included 6 studies and found weak to strong effect of neural gliding exercises. Recent studies have revealed complex nociceptive mechanisms involved in CTS which should be carefully considered during the management of these patients. Proper physical therapy interventions can modulate nociceptive processes found in CTS. We will perform a randomized clinical trial nested within a prospective cohort as our study design to determine if proper physical therapy approach targeted to modulate sensitization processes is equally effective than surgical intervention for improving pain and function in patients with carpal tunnel syndrome.

ELIGIBILITY:
Inclusion Criteria:

* pain and paresthesia in the median nerve distribution without extra-median nerve territory symptoms;
* increasing symptoms during night;
* Tinel sign;
* Phalen sign;
* self-reported hand strength deficits.
* Deficits of sensory and motor nerve conduction of the median nerve according to standardized guidelines of the American Association of Electrodiagnosis, American Academy of Neurology, and the American Academy of Physical Medicine and Rehabilitation

Exclusion Criteria:

* if any sensory/motor deficit in ulnar or radial nerve was present;
* previous interventions with surgery or steroid injections;
* multiple diagnoses of the upper extremity (i.e., cervical radiculopathy, lateral epicondylalgia);
* history of neck, shoulder or arm trauma;
* history of a systemic disease causing CTS (e.g. diabetes mellitus, or thyroid disease);
* history of systemic musculoskeletal conditions (e.g. rheumatoid arthritis, fibromyalgia);
* if the patient was actively involved with or seeking litigation at the time of the study;
* pregnancy.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-02-20 (Actual); Primary Completion 2014-01-25 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
Changes in the intensity of pain symptoms between baseline and follow-up periods | Baseline and 1, 3, 6 and 12 months after the intervention
  A 10-cm Numerical Pain Rating Scale(NPRS; 0: no pain, 10: maximum pain) will be used to assess current level of hand pain, and worst level of hand pain experienced in the preceding week.

SECONDARY OUTCOMES:
Changes in patients self-perceived improvement between baseline and follow-up periods | Baseline and 1, 3, 6 and 12 months after the intervention
  Patients self-perceived improvement will be assessed using a Global Rating of Change (GROC) consisting of a 15-point scale ranging from -7 (a very great deal worse) to +7 (a very great deal better). Descriptors of worsening or improving are assigned with values ranging from -1 to -7 and +1 to +7, respectively.
Changes in function between baseline and follow-up periods | Baseline, and 1, 3, 6 and 12 months after intervention
  The Spanish version of the Boston Carpal Tunnel Questionnaire (BCTQ) will be used. This questionnaire evaluates two domains: a) the functional status scale assesses ability to perform 8 common hand-related tasks; b) the symptom severity scale includes 11 items assessing pain severity, numbness, and weakness at night and during the day. Each question is answered on a 5 point scale (1: no complaint; 5: severe complaint), with higher scores indicating greater severity.
Changes in severity of the symptoms between baseline and follow-up periods | Baseline, and 1, 3, 6 and 12 months after the intervention
  The Spanish version of the Boston Carpal Tunnel Questionnaire (BCTQ) will be used. This questionnaire evaluates two domains: a) the functional status scale assesses ability to perform 8 common hand-related tasks; b) the symptom severity scale includes 11 items assessing pain severity, numbness, and weakness at night and during the day. Each question is answered on a 5 point scale (1: no complaint; 5: severe complaint), with higher scores indicating greater severity.

OTHER OUTCOMES:
Changes in Health-related quality of life (economic analysis) | Baseline, and 1, 3, 6 and 12 months after the intervention
  The paper-based five-level version of EuroQol-5D (EQ-5D-5L) was used.
Changes in the intensity of pain symptoms between baseline and 4 years follow-up (extended follow-up) | Baseline and 48 months after the intervention (extended follow-up)
  A 10-cm Numerical Pain Rating Scale(NPRS; 0: no pain, 10: maximum pain) will be used to assess current level of hand pain, and worst level of hand pain experienced in the preceding week.
Changes in function and severity of symptoms between baseline and 4 years follow-up (extended follow-up) | Baseline and 48 months after the intervention (extended follow-up)
  The Spanish version of the Boston Carpal Tunnel Questionnaire (BCTQ) will be used. This questionnaire evaluates two domains: a) the functional status scale assesses ability to perform 8 common hand-related tasks; b) the symptom severity scale includes 11 items assessing pain severity, numbness, and weakness at night and during the day. Each question is answered on a 5 point scale (1: no complaint; 5: severe complaint), with higher scores indicating greater severity.

CONTACTS AND LOCATIONS:
Overall Officials: César Fernández-de-las-Peñas, PT, PhD, DMSc, Principal Investigator — Universidad Rey Juan Carlos
Locations (1):
- Universidad Rey Juan Carlos - Hospital Universitario Fundación Alcorcon, Alcorcón, Madrid, Spain

REFERENCES:
- [Derived] Lopez-de-Uralde-Villanueva I, Fernandez-de-Las-Penas C, Cleland JA, Cook C, de-la-Llave-Rincon AI, Valera-Calero JA, Plaza-Manzano G. Minimal Clinically Important Differences in Hand Pain Intensity (Numerical Pain Rate Scale) and Related-Function (Boston Carpal Tunnel Questionnaire) in Women With Carpal Tunnel Syndrome. Arch Phys Med Rehabil. 2024 Jan;105(1):67-74. doi: 10.1016/j.apmr.2023.07.018. Epub 2023 Aug 13. PMID 37582474
- [Derived] Liew BXW, de-la-Llave-Rincon AI, Scutari M, Arias-Buria JL, Cook CE, Cleland J, Fernandez-de-Las-Penas C. Do Short-Term Effects Predict Long-Term Improvements in Women Who Receive Manual Therapy or Surgery for Carpal Tunnel Syndrome? A Bayesian Network Analysis of a Randomized Clinical Trial. Phys Ther. 2022 Apr 1;102(4):pzac015. doi: 10.1093/ptj/pzac015. PMID 35194646
- [Derived] Fernandez-de-Las-Penas C, Arias-Buria JL, Cleland JA, Pareja JA, Plaza-Manzano G, Ortega-Santiago R. Manual Therapy Versus Surgery for Carpal Tunnel Syndrome: 4-Year Follow-Up From a Randomized Controlled Trial. Phys Ther. 2020 Oct 30;100(11):1987-1996. doi: 10.1093/ptj/pzaa150. PMID 32766779
- [Derived] Fernandez-de-Las Penas C, Ortega-Santiago R, de la Llave-Rincon AI, Martinez-Perez A, Fahandezh-Saddi Diaz H, Martinez-Martin J, Pareja JA, Cuadrado-Perez ML. Manual Physical Therapy Versus Surgery for Carpal Tunnel Syndrome: A Randomized Parallel-Group Trial. J Pain. 2015 Nov;16(11):1087-94. doi: 10.1016/j.jpain.2015.07.012. Epub 2015 Aug 15. PMID 26281946